CLINICAL TRIAL: NCT01185015
Title: A Clinical Trial to Assess the Efficacy of Sigmart in Patients With Recurrent Angina After Coronary Revascularization
Brief Title: A Multi-centric Study to Assess the Efficacy of Sigmart in Subjects With Recurrent Angina After Coronary Revascularization
Acronym: SIGMART
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Cherry Ma, Beijing Merck Pharmaceutical Consulting LTD, an affiliate of Merck KGaA, Darmstadt, Germany.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200101-500
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2012-07

CONDITIONS: Angina Pectoris
Keywords: Angina Pectoris, Coronary disease
MeSH Terms: conditions — Angina Pectoris; Coronary Disease | interventions — Nicorandil

INTERVENTIONS:
Drug: Sigmart (nicorandil) — Sigmart will be administered for 2 weeks when the subject enters the secondary treatment period (Day 15 to approximately Day 28), at the dosage of 5 mg per oral tid in addition to the previous anti-anginal regimen.
  Other Names: Sigmart®

SUMMARY:
The multi-centric, open label, single arm and self controlled study is planned to assess the efficacy of orally administered Sigmart in subjects with recurrent angina after coronary revascularization. The primary objective of this study is to demonstrate that orally administered Sigmart can improve the major Exercise Tolerance Test (ETT) result in recurrent angina subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be 18~70 years old, male or female
* Subjects should have a history of coronary revascularization at least 6 months ago
* Subjects should present with typical angina or similar to the chest pain before prior coronary revascularization for at least 1 month
* Subjects should be relieved from anginal attacks with short-acting NTG
* Subjects should have the ability to withhold medication which cannot be concomitant in this clinical study during the study
* Subjects should have an ability to give written informed consent

Exclusion Criteria:

* Unstable angina
* Left main coronary artery disease
* Aortic stenosis
* Obstructive hypertrophic cardiomyopathy
* Subjects with hypertension (SBP>170 mmHg or DBP>100 mmHg) or hypotension (SBP<90 mmHg or DBP<60 mmHg)
* Postural hypotension (drop in systolic blood pressure >20% after 2 minute standing),
* Congestive heart failure (NYHA class III - IV)
* Ejection fraction (EF)<45% by Echocardiography
* Peripheral arterial obstructive disease or other diseases limiting exercise testing
* Arrhythmias requiring active treatment
* Gastro-intestinal ulcer
* Liver dysfunction (defined as ALT or bilirubin>1.5×upper limit of normal value)
* Significant renal impairment, such as serum creatinine greater than 1.5 folds the upper limit of normal as determined by local clinical laboratory
* Glaucoma
* Concomitant medication such as Trimetazidine, Sulphonylurea, PDE-5 inhibitor such as sildenafil, Chinese traditional medicine for treatment of angina pectoris
* Known intolerance to nitrates
* Known allergic to nicotinic acid
* Pregnant or lactating women
* Any other contraindications mentioned in the SPC
* Participation in another clinical study within the last 3 months
* Legal incapacity or limited legal capacity
* Any other subjects assessed by the investigator as being unsuitable for the present study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Time to 1 mm ST-depression | until day 28
  It is defined as the exercise time to develop 1 mm ST-segment depression in the same identified leads

SECONDARY OUTCOMES:
Exercise tolerance test parameters | until day 28
  Exercise Tolerance Test (ETT) parameters include:
  * Total exercise time
  * Time to onset of chest pain using ETT
  * Maximum ST-depression
  * SBP × HR (Pressure Rate Product)
  * Metabolic Equivalents (METs)
  * ETT grade and Score
Consumption of nitroglycerine (NTG). | until day 28
  Weekly assessment of NTG consumption until visit 4 (day 28)
Adverse events | until day 28
  The incidence of adverse events (especially the incidence of headache)
Compliance | until day 28
  Compliance % ([total number of tablets taken divided by the total number of tablets to be taken] multiplied by 100)
Number of angina attacks per week | until day 28
  Weekly assessment of angina attacks until day 28

CONTACTS AND LOCATIONS:
Overall Officials: Cherry Ma, PhD, Study Director — Beijing Merck Pharmaceutical Consulting Ltd., China